CLINICAL TRIAL: NCT01989169
Title: A Phase 1, Randomized, Open Label, Crossover Study to Evaluate the Pharmacokinetic Interaction Between SSP-004184 (SPD602) and Midazolam in Healthy Adult Subjects
Brief Title: Pharmacokinetic Interaction Between SSP-004184 (SPD602) and Midazolam in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPD602-117
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

ARMS (2):
- Midazolam (Active Comparator): Administered as a single oral 6 mg dose on Day 1.
  Interventions: Drug: Midazolam
- SSP-004184SS + Midazolam (Experimental): Midazolam (6 mg) + SSP-004184SS (30 mg/kg) concomitantly administered as a single oral dose on Day 1.
  Interventions: Drug: Midazolam; Drug: SSP-004184SS

INTERVENTIONS:
Drug: Midazolam
Drug: SSP-004184SS
  Other Names: SPD602
  Arms: SSP-004184SS + Midazolam

SUMMARY:
A Study to Evaluate the Pharmacokinetic Interaction Between SSP-004184 and Midazolam in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy male and female volunteers between the ages of 18 and 65, inclusive
* Serum ferritin, hemoglobin and erythrocyte indices within normal range

Exclusion Criteria:

* Evidence of any active or chronic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2014-01-06 (Actual); Study Completion 2014-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Midazolam First: Subjects received Midazolam 6mg in Period 1, followed by Midazolam 6mg and SSP-004184SS 30mg/kg during Period 2.
- Midazolam + SSP-004184SS First: Subjects received Midazolam 6mg and SSP-004184SS 30mg/kg in Period 1, followed by Midazolam 6mg during Period 2.
Period: Period 1
Arm/Group | Midazolam First | Midazolam + SSP-004184SS First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Midazolam First | Midazolam + SSP-004184SS First
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam First | Midazolam + SSP-004184SS First | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37 (10.45) | 44.9 (10.53) | 41 (11.07)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 14 | 15 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 11 | 10 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUCinf) of Midazolam
Description: AUCinf is the area under the plasma concentration versus time curve extrapolated from time 0 to infinity, calculated using the observed value of the last non-zero concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Study Periods 1 & 2: Within 60 minutes pre-dose, and Post-dose 0.167, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hours.
Population: Pharmacokinetic Set: All subjects who took at least 1 dose of investigational product and for whom the primary pharmacokinetic data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Midazolam | SSP-004184SS + Midazolam
Number analyzed (Participants) | 29 | 30
ng*hr/mL | 103.348 (54.087) | 120.1 (38.686)
Statistical Analysis 1: Comparison: Midazolam vs SSP-004184SS + Midazolam; The means of the log-transformed pharmacokinetic parameters were compared between treatments using a mixed-effects model with period and treatment as fixed effects and subject nested within sequence as a random effect. In order to estimate the magnitude of the treatment regimen differences in AUCinf, the geometric mean ratio (i.e., the least squares mean difference in the log-transformed parameters back transformed to the original scale) and their 90% CIs were calculated; Test type: Non-Inferiority or Equivalence — If the 90% CI of the geometric mean ratios were within the range (0.80, 1.25), then equivalence was assumed and the hypothesis that a drug interaction occurred was rejected. If the 90% CIs were not wholly contained within the range (0.80, 1.25), then a drug interaction was not excluded; Mixed-effects Model; Ratio of Geometric LS Means = 1.215, 90% CI 2-sided [1.116 to 1.323] — The ratio of geometric LS means and 90% CIs for the geometric mean ratio is for Treatment B to Treatment A

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measureable Concentration (AUClast) of Midazolam
Description: AUClast is the area under the concentration versus time curve from the time of dosing to the last measurable concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Midazolam | SSP-004184SS + Midazolam
Number analyzed (Participants) | 29 | 30
ng*h/ml | 100.935 (54.014) | 116.902 (37.45)
Statistical Analysis 1: Comparison: Midazolam vs SSP-004184SS + Midazolam; The means of the log-transformed pharmacokinetic parameters were compared between treatments using a mixed-effects model with period and treatment as fixed effects, and subject nested within sequence as a random effect. In order to estimate the magnitude of the treatment regimen differences in AUClast, the geometric mean ratio (i.e., the least squares mean difference in the log-transformed parameters back transformed to the original scale) and their 90% CIs were calculated; Test type: Non-Inferiority or Equivalence — If the 90% CI of the geometric mean ratios fell within the range (0.80, 1.25), then equivalence was assumed and the hypothesis that a drug interaction occurred was rejected. If the 90% CIs were not wholly contained within the range (0.80, 1.25), then a drug interaction was not excluded; Mixed-effects Model; Ratio of Geometric LS Means = 1.216, 90% CI 2-sided [1.115 to 1.327] — The ratio of geometric LS means and 90% CIs for the geometric mean ratio is for Treatment B to Treatment A

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Midazolam
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Midazolam | SSP-004184SS + Midazolam
Number analyzed (Participants) | 29 | 30
ng/mL | 35.124 (12.532) | 48.29 (12.605)
Statistical Analysis 1: Comparison: Midazolam vs SSP-004184SS + Midazolam; The means of the log-transformed pharmacokinetic parameters were compared between treatments using a mixed-effects model with period and treatment as fixed effects, and subject nested within sequence as a random effect. In order to estimate the magnitude of the treatment regimen differences in Cmax, the geometric mean ratio (i.e., the least squares mean difference in the log-transformed parameters back transformed to the original scale) and their 90% CIs were calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mixed-effects Model; Ratio of Geometric LS Means = 1.383, 90% CI 2-sided [1.282 to 1.491] — The ratio of geometric LS means and 90% CIs for the geometric mean ratio is for Treatment B to Treatment A

ADVERSE EVENTS:
Groups:
- Midazolam Alone: Administered as a single oral 20 mg dose on Day 1.
- Midazolam + SSP-004184SS: Midazolam (6 mg) + SSP-004184SS (30 mg/kg) administered concomitantly as a single oral dose on Day 1.
Arm/Group | Midazolam Alone | Midazolam + SSP-004184SS
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 6/29 | 10/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam Alone (N=29) | Midazolam + SSP-004184SS (N=30)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5)
Somnolence (Nervous system disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.